CLINICAL TRIAL: NCT04773730
Title: A Comparative Study Between Quadratus Lumborum Block Type 2 and Posterior Transversus Abdominus Plane Block for Analgesia After Cesarean Delivery Under Spinal Anesthesia
Brief Title: Quadratus Lumborum Block Type 2 Versus Posterior Transversus Abdominus Plane Block
Acronym: quadratus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, maha abou-zeid, Assistant professor of anesthesia and surgical intensive care, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: regional block
Record Dates: First submitted 2021-02-20; First posted 2021-02-26 (Actual); Last update posted 2023-06-06 (Actual); Status verified 2023-06

CONDITIONS: Regional Block

STUDY DESIGN:
Intervention Model Description: patients will be randomly allocated via sealed opaque envelop into 2 groups of 50 patients each; Posterior transversus abdominus block (TAP) group and Quadratus lumborum block type 2 is the second group (QLB)group
Who Masked: Participant, Investigator
Masking Description: pain score assessment will be done by an anesthetist who is not involved in randomization or in the anesthetic technique
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Posterior transversus abdominus block (Active Comparator): After the surgery end and while the patient in the supine position, with the side to be blocked is elevated
  A 12-14 MHz linear array transducer will be placed transversely between the iliac crest and costal margin then slided from medial-lateral to visualize the posterior most part of the external oblique, internal oblique, and transversus abdominus muscles
  Then 20 mL of bupivacaine0.25% will be injected between the transverses abdominus muscle and the fascia deep to the internal oblique muscle
  The same steps will be repeated on the other side
  Interventions: Procedure: Posterior transversus abdominus plane block
- Quadratus lumborum block type 2 (Active Comparator): After the surgery end and while the patient in the supine position, with the side to be blocked is elevated
  A2-5 MHz curved array transducer will be placed at the level of the antero-superior iliac spine then the external oblique muscle will be followed posterolaterally until its posterior border will be visualized The probe will be tilted down to identify a bright hyperechoic line After that 20 mL of bupivacaine 0.25% will be injected under direct visualization on the posterior surface of quadrates lumborum muscle
  The same steps will be repeated on the other side
  Interventions: Procedure: Quadratus lumborum block type 2

INTERVENTIONS:
Procedure: Posterior transversus abdominus plane block — Twenty mL of bupivacaine 0.25% will be injected in the plane between the transverses abdominus muscle and the fascia deep to the internal oblique muscle on each side
  Arms: Posterior transversus abdominus block
Procedure: Quadratus lumborum block type 2 — Twenty mL of bupivacaine 0.25% will be injected on the posterior surface of quadrates lumborum muscle on each side
  Arms: Quadratus lumborum block type 2

SUMMARY:
This patient population are at risk of adverse effects secondary to inadequate pain management such as inadequate maternal bonding and late ambulation.

Regional analgesia is preferred due to their opioid sparing effects and reduction in related adverse effects but the analgesia from these blocks is not known which one is superior to the other in the context of cesarean section

DETAILED DESCRIPTION:
The aim of this study is to compare the effect of posterior transversus abdominus plane block and quadratus lumborum type 2 for cesarean delivery.

The transversus abdominus plane(TAP) block provides sensory block from T6 to L1 for lower abdominal surgeries.

Quadratous lumborum type 2 block, the injection is posterior to the quadratus lumborum muscle. This method has the advantage of a more superficial point of injection with better ultrasonographic resolution.

Only one RCT was done in this context by Kalpana Verma and his colleagues comparing quadratus lumborum type 2 and posterior transversus abdominus plane block. That shows marked discrepancy with time to first analgesic request from the quadratus lumborum block in other abdominal surgeries

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical status II parturient.
* Singleton pregnancies with a gestation of at least 37 weeks.
* Patients undergoing spinal anesthesia for cesarean deliveryvia a Pfannenstiel incision with exteriorization of the uterus.

Exclusion Criteria:

* Age < 19 or > 40 years.
* Height<150 cm, weight < 60 kg, body mass index (BMI) ≥35 kg/m2.
* Inability to comprehend or participatein pain scoring system.
* Contraindications to spinal anesthesia (Coagulopathy, increased intracranial pressure, or local skin infection).
* Hypersensitivity to any drugused in the study.
* Hypertensive disorders of pregnancy.
* Renal impairment or other contraindication to non-steroidal anti-inflammatory drugs.
* Significant cardiovascular, renal or hepatic abnormalities.
* Patients with history of opoid intake, drug abusers, psychiatric patients.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Parturient Female patients
Enrollment: 100 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2023-06-03 (Actual)

PRIMARY OUTCOMES:
The analgesic duration | within 24 hours after the surgery
  the time measured from finishing the block till the first request of analgesia by the patient

SECONDARY OUTCOMES:
Postoperative pain at rest | immediately and 1,2,3,4hour at postanesthesia care unit, then in the surgical ward at 6,8,10,12,18 and 24 h
  100 centimetres visual analog scale (VAS) for pain, where zero is equal to no pain and hundred indicates the worst possible pain
Postoperative pain on movement (attempted hip flexion) or coughing | immediately and 1,2,3,4hour at postanesthesia care unit, then in the surgical ward at 6,8,10,12,18 and 24 h
  100 centimetres visual analog scale (VAS) for pain, where zero is equal to no pain and hundred indicates the worst possible pain
Patient satisfaction | 24 hours after surgery
  poor= 1, fair = 2, good = 3, excellent = 4
Heart rate | at 1st, 2nd, 3rd, 4th, 10th, 16th and 22nd hours postoperatively
  beat per minute
Non-invasive blood pressure | at 1st, 2nd, 3rd, 4th, 10th, 16th and 22nd hours postoperatively
  mmHg
Total postoperative analgesic consumption of of ketolac, paracetamol and fentanyl | within the first 24 hours after surgery
  Patients with visual analog scale more than 30 will receive 30 mg of intravenous ketolac in addition to 1gm paracetamol which will be repeated every 8 hours intravenous infusion of every 8 hours. Intravenous administration of fentanyl bolus doses of 0.5 µg per kg per dose will be given if the visual analog scale remains more than 30
Postoperative nausea and vomiting | within 24 hours after surgery
  0= none, 1= mild, 2= moderate and 3= sever
Postoperative lower limb weakness | within 24 hours after surgery
  reported by the patient during her first walk after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Maha Ahmed Abozeid, MD, Study Director — Faculty of Medicine - Mansoura University
Locations (1):
- El Mansoura, El Mansoura, Egypt